CLINICAL TRIAL: NCT01685398
Title: Treatment of Cutaneous Hemangioma of Infancy With Topical 0.5% Timolol Maleate Eye Drop Compared With Placebo in Pediatric Patients, Siriraj Hospital
Brief Title: Topical Timolol for Superficial Infantile Hemangioma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 088/2555(EC4)
Record Dates: First submitted 2012-09-05; First posted 2012-09-14 (Estimated); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Hemangioma
MeSH Terms: conditions — Hemangioma | interventions — Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- normal saline (Placebo Comparator): normal saline 1-2 drops put on the hemangioma lesion 4 times a day and rub over the entire lesion with a finger
  Interventions: Drug: Normal saline
- 0.5% timolol maleate eye drop (Experimental): 0.5% timolol maleate solution 1-2 drops put on the hemangioma lesion 4 times a day and rub over the entire lesion with a finger
  Interventions: Drug: 0.5% timolol maleate eye drop

INTERVENTIONS:
Drug: 0.5% timolol maleate eye drop
  Arms: 0.5% timolol maleate eye drop
Drug: Normal saline
  Other Names: Saline
  Arms: normal saline

SUMMARY:
Infantile hemangioma (IH) is the most common benign vascular tumor in pediatric population. The characteristic natural history of this tumor is rapid growth in the first year of life and follows by spontaneous involution. However, it may cause cosmetic unacceptable. Early intervention in superficial IH may help to minimize the risk of residual aesthetic problems. Topical timolol, a non selective beta-blocker, is an emerging treatment which has been reported in efficacy and safety for the treatment of IH. However, the reported studies were case-series or small study. This study is a prospective double-blind,randomized-controlled study to evaluate the efficacy and safety of 0.5% timolol maleate solution for treatment in superficial IH. The patient will be treated with topical timolol for at least 6 months and instructed to 4 times daily apply 1-2 drop of timolol solution on the lesion and rub over the entire lesion with a finger. Photographs of the lesion will be taken at the baseline and every 1-month visit. Clinical evaluation of the treatment efficacy is carried out by 2 investigators independently to determine the change in lesion size and visual analogue scale of the lesion color. The main outcome is to evaluate the efficacy of 0.5% timolol maleate solution in treatment of infantile hemangioma compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patient who is less than 2 years
* Patient who has been diagnosed with superficial infantile hemangioma
* The tumor which has been in proliferative or plateau phase
* There is no indication for systemic treatment
* Informed consent is obtained from the parent of the patient

Exclusion Criteria:

* Patient who has the indication for systemic therapy
* Patient who is treated by the other modality such as laser treatment
* Patient who has underlying disease treated by beta blocker, corticosteroids, interferon, cyclophosphamide or vincristine
* Patient who has history of hypersensitivity reaction to beta blocker, asthma, cardiac condition prove to heart block

Max Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2023-03 (Actual); Study Completion 2023-03 (Actual)

PRIMARY OUTCOMES:
Efficacy of the topical 0.5% timolol maleate solution in treatment of infantile hemangioma compared to placebo | 6 months
  Percent changes in visual analogue scale of the lesion color and global assessment scale of the lesion after treatment

SECONDARY OUTCOMES:
Side effects of the topical 0.5% timolol maleate solution in treatment of infantile hemangioma | 6 months
  The side effects of 0.5% timolol maleate solution include bradycardia, dizziness, irritant contact dermatitis, allergic contact dermatitis, fatigue, nausea, diarrhea,and insomnia. To determine the side effects, investigators will monitor the vital signs of the patients every follow-up visit and ask the caretakers about the side effects. Furthermore, every patients will receive the dairy to record the frequency of drug usage and side effects found.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Siriraj Hospital Mahidol University, Bangkoknoi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No